CLINICAL TRIAL: NCT01629680
Title: A Randomized, Placebo-controlled Study Investigating the Effects of Moxaverine on Ocular Blood Flow After Oral Administration in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Associate Prof. PD Dr, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-080210
Record Dates: First submitted 2012-06-11; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Effect of Orally Administrated Moxaverine on Ocular Blood Flow
Keywords: moxaverine; ocular blood flow
MeSH Terms: interventions — moxaverine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy subjects I (Experimental)
  Interventions: Drug: Moxaverine
- Healthy subjects II (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxaverine — Moxaverine-hydrochloride, coated tablets containing 150 mg moxaverine (Kollateral forte, Ursapharm. Saarbrücken, Germany), dosage: 900 mg, administrated per os in three equal doses of 300 mg at two hour intervals
  Arms: Healthy subjects I
Drug: Placebo — coated tablets identical in number and appearance as the study drug
  Arms: Healthy subjects II

SUMMARY:
A number of common eye diseases such as age-related macular degeneration and glaucoma are associated with ocular perfusion abnormalities. Although this is well recognized there is not much possibility to improve blood flow to the posterior pole of the eye in these diseases.

For many years, moxaverine has been used in the therapy of perfusion abnormalities in the brain, the heart and the extremities. This is based on a direct vasodilatatory effect of the drug, but also on the rheological properties of red blood cells. In two recent studies the investigators have shown that intravenous moxaverine increases choroidal and retrobulbar blood flow in healthy young subjects, in elderly people with healthy eyes and in patients with eye diseases associated with hypoperfusion. The present study aims to investigate, whether ocular blood flow is also improved after oral administration of moxaverine.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmoker
* Body mass index between 16 and 30 kg/m²
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 dpt, anisometropia < 2 dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages or drugs
* Participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of the study drug
* Blood donation during the previous 3 weeks
* Presence of any ocular pathology that interferes with the aims of the present study
* Hypersensitivity to moxaverine
* Acute gastric bleeding, massive cerebral hemorrhage related to stroke
* Women: pregnancy or lactation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Choroidal and optic nerve head blood flow | 2 weeks
  Change in choroidal and optic nerve head blood flow after administration of moxaverine compared to placebo (measured before administration and 6 hours after administration)

SECONDARY OUTCOMES:
Retrobulbar flow velocities | 2 weeks
  Change in retrobulbar flow velocities after administration of moxaverine compared to placebo (measured before administration and 6 hours after administration)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria